CLINICAL TRIAL: NCT04370080
Title: Silver Diamine Fluoride Treatment of Active Root Caries Lesions in Older Adults: A Case Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roseman University of Health Sciences (Other)
Responsible Party: Principal Investigator, David Prince, Associate Professor, Roseman University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1122117-4
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Root Caries
MeSH Terms: conditions — Root Caries

STUDY DESIGN:
Intervention Model Description: Case series, consecutive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Silver Diamine Fluoride (Experimental): Topical application of one drop of silver diamine fluoride 38% to active untreated roof surface caries, lesions at the furcation, or lesions at crown margins. Application was repeated once each six months.
  Interventions: Device: Silver Diamine Fluoride 38%

INTERVENTIONS:
Device: Silver Diamine Fluoride 38% — Dental caries arrest medication
  Other Names: Advantage Silver Arrest

SUMMARY:
The authors conducted a case series to determine the outcomes of treatment of root surface caries lesions when the teeth were treated topically with 38% silver diamine fluoride.

DETAILED DESCRIPTION:
The study is a prospective, single center case series. The cases were consecutive. Participation was offered to every patient who qualified based on age and the presence of an active lesion in a root surfaces, in a furcation, or under an individual crown or crown abutment for a fixed prosthesis. The study was conducted at the dental clinic of the Roseman College of Dental Medicine in South Jordan, Utah. The University of California, San Francisco protocol for applying topical silver diamine fluoride was adapted for use with these patients. Lesions were flushed with water and then dried with compressed air, isolated with cotton rolls, and then 38% silver diamine fluoride (Advantage Arrest, Elevate Oral Care, West Palm Beach, FL) was applied repeatedly for two minutes with the manufacturer supplied dental applicator. The silver diamine fluoride was stored under the manufacturer's recommended conditions. If the patient complained about the taste, the lesion was coated with sodium fluoride varnish. All of the lesions were reevaluated for dental caries lesion activity about every six months and retreated regardless of their arrest status. Follow-up was for 30 months or until loss to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 active root surface caries lesion by Nyvad criteria

Exclusion Criteria:

* None

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Dental caries lesion activity 1 | 6-12 months
  Nyvad score based on visual/tactile examination
Dental caries lesion activity 2 | <6 months
  Nyvad score based on visual/tactile examination
Dental caries lesion activity 3 | 12-18 months
  Nyvad score based on visual/tactile examination
Dental caries lesion activity 4 | 18-24 months
  Nyvad score based on visual/tactile examination
Dental caries lesion activity 5 | 24-30 months
  Nyvad score based on visual/tactile examination

SECONDARY OUTCOMES:
Caries lesion fluorescence 1 | <6 months
  Laser fluorescence measurement at the surface of the lesion
Caries lesion fluorescence 2 | 6-12 months
  Laser fluorescence measurement at the surface of the lesion
Caries lesion fluorescence 3 | 12-18 months
  Laser fluorescence measurement at the surface of the lesion
Caries lesion fluorescence 4 | 18-24 months
  Laser fluorescence measurement at the surface of the lesion
Caries lesion fluorescence 5 | 24-30 months
  Laser fluorescence measurement at the surface of the lesion

CONTACTS AND LOCATIONS:
Overall Officials: David Prince, DDS, Principal Investigator — Roseman Health Sciences University

REFERENCES:
- [Background] Nyvad B, Machiulskiene V, Baelum V. Reliability of a new caries diagnostic system differentiating between active and inactive caries lesions. Caries Res. 1999 Jul-Aug;33(4):252-60. doi: 10.1159/000016526. PMID 10343087
- [Derived] Mitchell C, Gross AJ, Milgrom P, Mancl L, Prince DB. Silver diamine fluoride treatment of active root caries lesions in older adults: A case series. J Dent. 2021 Feb;105:103561. doi: 10.1016/j.jdent.2020.103561. Epub 2020 Dec 24. PMID 33347946